CLINICAL TRIAL: NCT05083572
Title: Effect of Probiotic (Vivomixx/ DeSimone Formulation) on Gut Microbiome and Bacterial Translocation in Healthy Asian Volunteers - An Exploratory Randomized Controlled Trial
Brief Title: Effect of Probiotic on Gut Microbiome and Bacterial Translocation in Healthy Asian Volunteers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Tiing Leong Ang, Chief and Senior Consultant, Department of Gastroenterology and Hepatology, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vivomixx
Record Dates: First submitted 2021-10-03; First posted 2021-10-19 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Dysbiosis
Keywords: Gut microbiome; Probiotic; Bacterial translocation
MeSH Terms: conditions — Dysbiosis | interventions — Polyethylene Glycols; Probiotics; Anti-Bacterial Agents; Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This will be a randomized controlled, partially-blinded study with four study arms to (i) examine the effect of Vivomixx on the gut microbiome with and without colonic lavage, (ii) with and without antibiotic treatment, (iii) compare the gut microbiome after natural recovery and with Vivomixx treatment following colonic lavage, and (iv) evaluate the efficacy of Vivomixx in reducing bacterial translocation and oxidative stress. The subjects will not be informed of the identity of the study product (Vivomixx or placebo) given. However, it is not possible to blind the subjects of the colonic lavage and rifaximin interventions. The investigators and outcomes assessors involved in the data analysis will be blinded to the study group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Lavage and Vivomixx) (Experimental): Colonic lavage, followed by Vivomixx treatment
  Interventions: Drug: Colonic lavage with polyethylene glycol; Dietary Supplement: Probiotic
- Group B (Lavage and Placebo) (Experimental): Colonic lavage, followed by Placebo treatment
  Interventions: Drug: Colonic lavage with polyethylene glycol
- Group C (Vivomixx) (Experimental): No colonic lavage, only Vivomixx treatment
  Interventions: Dietary Supplement: Probiotic
- Group D (Rifaximin and Vivomixx) (Experimental): Rifaximin, followed by Vivomixx treatment
  Interventions: Dietary Supplement: Probiotic; Drug: Antibiotic

INTERVENTIONS:
Drug: Colonic lavage with polyethylene glycol — The subjects will orally consume a split dose of bowel preparation (PEG); 2 litres in the evening (Day -1) and another 2 litres the following morning (Day 1).
  Other Names: PEG
  Arms: Group A (Lavage and Vivomixx); Group B (Lavage and Placebo)
Dietary Supplement: Probiotic — The subjects will self-administer orally two capsules of Vivomixx with room temperature water (as heat may inactivate the live bacteria, rendering it less effective) twice daily for 28 days.
  Other Names: Vivomixx
  Arms: Group A (Lavage and Vivomixx); Group C (Vivomixx); Group D (Rifaximin and Vivomixx)
Drug: Antibiotic — The subjects will undergo pre-treatment to "cleanse" the gut by consuming orally one tablet of antibiotic rifaximin (200mg) daily for 14 days prior to the initiation of Vivomixx course.
  Other Names: Rifaximin
  Arms: Group D (Rifaximin and Vivomixx)

SUMMARY:
Dysbiosis of the gut microbiome has been recognized to underlie the pathogenesis of various gastrointestinal conditions. Probiotics are known to exert beneficial effects on gut health and have great potential for use as microbiome interventions for gastrointestinal and metabolic diseases. While it is widely known that probiotic bacteria favourably alter the intestinal microflora balance, their other mechanisms of action have not been systematically characterized. The ability of probiotics to modulate dysbiosis may lead to reduced levels of endotoxaemia and oxidative stress. In this study, the investigators propose to examine the effects of 4-week Vivomixx treatment on the gut microbiome and bacterial translocation in healthy Asian volunteers with and without colonic lavage or antibiotic treatment. The study will also examine the same outcome parameters 4 weeks upon cessation of the product. The findings derived from the study will provide valuable insights into the microbiota changes associated with colonic lavage or antibiotic treatment, and the use of probiotic (Vivomixx). This has important clinical implications in designing treatment strategies in clinical practice such as the use of Vivomixx as microbiome interventions with antibiotics which are known to induce Clostridium difficile-associated diarrhoea, as well as in the therapeutic management of various diseases associated with dysbiosis.

DETAILED DESCRIPTION:
This will be a randomized controlled, partially-blinded study with four study arms to (i) examine the effect of Vivomixx on the gut microbiome with and without colonic lavage, (ii) with and without antibiotic treatment, (iii) compare the gut microbiome after natural recovery and with Vivomixx treatment following colonic lavage, and (iv) evaluate the efficacy of Vivomixx in reducing bacterial translocation and oxidative stress.

Screening Visit Procedures (within 28 days of first dosing):

* Informed consent;
* Demography, including date of birth, sex, and race/ethnicity;
* Body weight and height measurement;
* Determination of eligibility based on inclusion/exclusion criteria;
* Adverse event/concomitant medication check;
* Complete medical/drug history;
* Alcohol/Smoking history;
* Blood pressure, heart rate and temperature, taken after resting at a sitting position for at least 5 minutes;
* Complete physical examination;
* Laboratory safety tests (liver panel, renal panel and complete blood count) (10 ml blood);
* Urine dipstick pregnancy test (for female subjects only).

Day -14 Procedures (for Group D only):

On reporting to CTRU on Day -14, participants will be reminded of study restrictions and undergo the following assessments:

* Interim medical/drug history;
* Adverse event/concomitant medication check;
* Blood pressure, heart rate and temperature, taken after resting at a sitting position for at least 5 minutes;
* Complete physical examination;
* Provision of baseline stool sample ~3g (before dosing with rifaximin) (for microbiome and SCFA);
* Provision of baseline blood sample ~12ml for flow cytometry and SCFA analysis (before dosing with rifaximin);
* Rifaximin on-site dosing;
* Rifaximin dispensing for home consumption (1 tablet 200mg daily till Day -7).

Day -7 Procedures (for Group D only):

On reporting to CTRU on Day -7, participants will be reminded of study restrictions and undergo the following assessments:

* Interim medical/drug history;
* Adverse event/concomitant medication check;
* Blood pressure, heart rate and temperature, taken after resting at a sitting position for at least 5 minutes;
* Brief physical examination;
* Provision of stool sample ~3g (for microbiome and SCFA);
* Provision of blood sample ~12ml for flow cytometry and SCFA analysis;
* Rifaximin home dosing (1 tablet 200mg in morning);
* Return of rifaximin for accountability check;
* Rifaximin dispensing for home consumption (1 tablet 200mg daily till Day 1).

Day -1 Procedures (for Groups A & B only):

On reporting to CTRU on Day -1, participants will be reminded of study restrictions and undergo the following assessments:

* Interim medical/drug history;
* Adverse event/concomitant medication check;
* Blood pressure, heart rate and temperature, taken after resting at a sitting position for at least 5 minutes;
* Complete physical examination;
* Provision of baseline stool sample ~3g (before dosing with PEG) (for microbiome and SCFA);
* Provision of baseline blood sample ~12ml for flow cytometry and SCFA analysis (before dosing with PEG);
* PEG dispensing for colonic lavage (home consumption- 2L at 6pm);
* Telephone call at night for bowel movement and AE check.

Day 1 Procedures:

• Home consumption of 2L PEG at 6am for colonic lavage.

On reporting to CTRU on Day 1, participants will be reminded of study restrictions and undergo the following assessments:

* Interim medical/drug history (for Group C only);
* Adverse event/concomitant medication check;
* Blood pressure, heart rate and temperature, taken after resting at a sitting position for at least 5 minutes (for Group C only);
* Complete physical examination;
* Verbal stool symptom assessment (for Group D only);
* Laboratory safety tests (liver panel, renal panel and complete blood count) (10 ml blood) (for Group D only);
* Biomarker test (5 ml blood before dosing) (for Group C only);
* Endotoxaemia test (5 ml blood 2hrs post-meal) (for Group C only);
* Provision of stool sample ~3g (before dosing with Vivomixx or Placebo) (for microbiome and SCFA);
* Provision of blood sample ~12ml for flow cytometry and SCFA analysis (before dosing with Vivomixx or Placebo);
* Vivomixx (Groups A, C & D) or Placebo (Group B) on-site dosing;
* Return of PEG (Groups A & B) or rifaximin (Group D) for accountability check;
* Vivomixx or Placebo dispensing for home consumption.

Day 2-28 Procedures:

* Self-administration of 2 capsules of Vivomixx (Groups A, C & D) or Placebo (Group B) twice daily (morning and evening) till Day 28;
* Consumption of the study products will be monitored real-time via electronic means on mobile devices (video call). All morning dosing should be between 8-10am, and all evening dosing should happen between 6-8pm;
* Verbal stool symptom assessment on Day 14.

Day 29 Procedures (+ 2 days):

On reporting to CTRU on Day 29, participants will be reminded of study restrictions and undergo the following assessments:

* Adverse event/concomitant medication check;
* Blood pressure, heart rate and temperature, taken after resting at a sitting position for at least 5 minutes;
* Verbal stool symptom assessment;
* Complete physical examination;
* Laboratory safety tests (liver panel, renal panel and complete blood count) (10 ml blood);
* Biomarker and endotoxaemia tests (10 ml blood) (for Group C only);
* Provision of stool sample ~3g (for microbiome and SCFA);
* Provision of blood sample ~12ml for flow cytometry and SCFA analysis;
* Vivomixx (Groups A, C & D) or Placebo (Group B) home dosing (2 capsules in morning and evening);
* Return of Vivomixx (Groups A, C & D) or Placebo (Group B) for accountability check.

Day 56 Procedures (± 3 days) (Final Visit):

* Adverse event/concomitant medication check;
* Brief physical examination;
* Verbal stool symptom assessment;
* Provision of stool sample ~3g (for microbiome and SCFA);
* Provision of blood sample ~12ml for flow cytometry and SCFA analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent,
2. Aged between 21-65 years of age,
3. Chinese, Malay or Indian ancestry through three generations,
4. Body Weight ≥ 50kg, Body Mass Index (BMI) of 18.5 to 29.9 kg/m2, inclusive,
5. Clinical laboratory assessment results within normal limits, unless the deviation is considered not clinically significant by the investigator,
6. Regular stool every 1-2 days,
7. Satisfactory medical assessment as assessed by physical examination, medical history, and normal laboratory values or minor variations that are not clinically significant,
8. Ability to communicate with the investigator and to understand and comply with all requirements of study participation.
9. Both male and female participants (with child-bearing potential) and their partners have to practise contraception throughout the duration of the study.

Exclusion Criteria:

1. Any acute illness within 14 days of first dosing, unless otherwise approved by the PI,
2. History or evidence of clinically significant hepatic, renal, cardiovascular, respiratory, gastrointestinal, immunosuppressive or metabolic disorders, any cancer types,
3. Declare themselves positive for HIV or viral hepatitis (Hepatitis A, B, C),
4. Treatment within the previous 3 months with antibiotics (subjects are to inform study staff should they be prescribed antibiotics during the course of the study)
5. Treatment with any prescription or over-the-counter medications, complementary health products, or herbal supplements within 28 days of first dosing,
6. Consumption of probiotics or lactobacillus-containing products e.g. Yakult, Vitagen or Yogurt within 4 weeks of first dosing unless approved by the PI,
7. Abnormal biochemistry indicators, unless certified as not clinically significant,
8. Poor peripheral venous access,
9. Irregular bowel habits or complains of constipation problem,
10. Pregnancy or lactation,
11. Known allergic reactions to rifaximin, PEG or Vivomixx,
12. History of drug/alcohol abuse,
13. Involvement in the planning or conduct of this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Microbiome profile using 16S rRNA sequencing | 2 to 2.5 months
  Fresh stool samples will be collected for microbial DNA extraction at Days -14 and -7 (Group D), Day -1 (Groups A & B), Days 1, 29 and 56 (All groups). Microbial DNA will be extracted from the stool samples and used for 16S rRNA sequencing. Bacterial species present in Vivomixx will be specifically examined.
Inflammatory cytokines using ELISA tests | 2 to 2.5 months
  Inflammatory cytokines indicative of oxidative damage will be assayed using commercially available Elisa kits on serum samples obtained at Baseline and Day 29 (For Group C only).
Bacterial translocation using endotoxin assay | 2 to 2.5 months
  Blood will be collected 2 hours post meal at baseline and Day 29 for endotoxin LAL assay using commercial kit (For Group C only).

SECONDARY OUTCOMES:
Peripheral blood lymphocyte phenotyping using flow cytometry | 2 to 2.5 months
  Blood will be collected at specified timepoints for peripheral blood lymphocyte phenotyping by flow cytometry
Short chain fatty acids using mass spectrometry | 2 to 2.5 months
  Stool and blood will be collected at specified timepoints for short chain fatty acid analysis by gas chromatography-mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Tiing Leong Ang, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jalanka J, Salonen A, Salojarvi J, Ritari J, Immonen O, Marciani L, Gowland P, Hoad C, Garsed K, Lam C, Palva A, Spiller RC, de Vos WM. Effects of bowel cleansing on the intestinal microbiota. Gut. 2015 Oct;64(10):1562-8. doi: 10.1136/gutjnl-2014-307240. Epub 2014 Dec 19. PMID 25527456
- [Background] Valentini L, Pinto A, Bourdel-Marchasson I, Ostan R, Brigidi P, Turroni S, Hrelia S, Hrelia P, Bereswill S, Fischer A, Leoncini E, Malaguti M, Blanc-Bisson C, Durrieu J, Spazzafumo L, Buccolini F, Pryen F, Donini LM, Franceschi C, Lochs H. Impact of personalized diet and probiotic supplementation on inflammation, nutritional parameters and intestinal microbiota - The "RISTOMED project": Randomized controlled trial in healthy older people. Clin Nutr. 2015 Aug;34(4):593-602. doi: 10.1016/j.clnu.2014.09.023. Epub 2014 Oct 8. PMID 25453395